CLINICAL TRIAL: NCT01601041
Title: Role of Residual Urine and Asymptomatic Prostatitis in the Development of Lower Urinary Tract Infections in Spinal Cord Injury Patients - a Prospective Study
Brief Title: Role of Residual Urine and Asymptomatic Prostatitis in the Development of Urinary Tract Infections in Spinal Cord Injury
Status: Completed | Type: Observational
Sponsor: Swiss Paraplegic Research, Nottwil (Network)
Responsible Party: Sponsor
Other Study IDs: 2011-16
Record Dates: First submitted 2012-05-01; First posted 2012-05-17 (Estimated); Last update posted 2016-11-22 (Estimated); Status verified 2016-11

CONDITIONS: Urinary Tract Infection
Keywords: Urinary Tract Infection; Bacteriuria; Pyuria; Prostatitis; Intermittent Catheterization; Spinal Cord Injuries; Residual Urine
MeSH Terms: conditions — Urinary Tract Infections; Bacteriuria; Pyuria; Prostatitis; Spinal Cord Injuries | interventions — High-Energy Shock Waves; Intermittent Urethral Catheterization

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- urinary tract infection: urinary tract infection in male patients with neurogenic bladder dysfunction due to spinal cord injury managed by intermittent catheterization
  Interventions: Other: sonographic assessment of residual urine, urine culture
- control group: less than three urinary tract infections / year
  Interventions: Other: sonographic assessment of residual urine, urine culture

INTERVENTIONS:
Other: sonographic assessment of residual urine, urine culture — residual urinary volume assessed by ultrasound after bladder catheterization urinary cultures taken before and after prostate massage
  Other Names: ultrasound; intermittent catheterization

SUMMARY:
The purpose of this prospective study is to investigate the association between the amount of residual urine and asymptomatic bacterial prostate infection with the occurrence of recurrent (>2 /year) symptomatic urinary tract infections in patients suffering from chronic (> 1 year) spinal cord injury (SCI) and neurogenic lower urinary tract dysfunction performing intermittent catheterization.

The following hypotheses will be tested:

1. The amount of residual urine after intermittent catheterization is significantly greater in SCI patients suffering from frequent (>2 /year) urinary tract infections compared to those without.
2. The incidence of asymptomatic bacterial prostate infections is significantly higher in SCI patients suffering from frequent (>2 /year) urinary tract infections compared to those without.

DETAILED DESCRIPTION:
To investigate the association between the amount of residual urine and asymptomatic bacterial prostate infection with the occurrence of recurrent (>2 /year) symptomatic urinary tract infections in patients suffering from chronic (> 1 year) spinal cord injury (SCI) and neurogenic lower urinary tract dysfunction performing intermittent catheterization, patients perform self-catheterization twice (before and after urodynamic testing. After each catheterization, residual urine is assessed by ultrasound. Prior to urodynamic testing, prostate massage is performed, bacterial cultures of the fluid and the urine are initiated and the results of these cultures will be analysed .

ELIGIBILITY:
Inclusion Criteria:

* male patients with chronic (> 1 year) spinal cord injury
* bladder management by intermittent catheterization

Exclusion Criteria:

* symptomatic urinary tract infection
* prostate pathology
* immunodeficiency
* antibiotic therapy
* missing informed consent

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male patients with chronic (> 1 year) spinal cord injury who perform intermittent catheterization due to neurogenic bladder dysfunction
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2011-12; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
amount of residual urine | change from self-catheterization 10 minutes before and 10 minutes after urodynamic assessment
  determined by ultrasound

SECONDARY OUTCOMES:
bacterial prostate infection | 5-10 minutes before and after prostate massage
  urinary culture
bacteriuria | 5-10 minutes before and after prostate massage
  urine dip stick
number of leucocytes in urine | 5-10 minutes before and after prostate massage
  urine dip stick
number of erythrocytes in urine | 5-10 minutes before and after prostate massage
  urine dip stick
patient characteristics | day 0
  age
type of neurogenic bladder dysfunction | day 0
type of catheter used for intermittent catheterization | day 0
annual rate of symptomatic urinary tract infections | day 0
patient characteristics | day 0
  sex
patient characteristics | day 0
  time since spinal cord injury
patient characteristics | day 0
  level and degree of spinal cord injury (ASIA impairment score)

CONTACTS AND LOCATIONS:
Overall Officials: Jürgen Pannek, Prof., Principal Investigator — Swiss Paraplegic Center, Nottwil, Switzerland
Locations (1):
- Swiss Paraplegic Centre, Nottwil, Canton of Lucerne, Switzerland